CLINICAL TRIAL: NCT01300039
Title: Oral Antibiotic Treatment of Helicobacter Pylori Reduces Intestinal Colonization Rates With Oxalobacter Formigenes
Status: Completed | Type: Observational
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: David S Goldfarb MD, New York Harbor VA Medical Center
Other Study IDs: 573
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Nephrolithiasis
Keywords: nephrolithiasis; urolithiasis; hyperoxaluria; Helicobacter pylori
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis; Hyperoxaluria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Antibiotics for H. pylori: Patients who underwent upper endoscopy and were found to have H. pylori, and were then to be treated with antibiotics for eradication of H. pylori
- Control group, no H. pylori: Patients who underwent upper endoscopy and found to not have H. pylori, and then would not receive antibiotics

SUMMARY:
The investigators are finding out if giving antibiotics for Helicobacter pylori will eliminate colonization of the colon by Oxalobacter formigenes.

DETAILED DESCRIPTION:
Background and objectives: Oxalobacter formigenes (OF) may play a protective role in preventing calcium oxalate stones. Intestinal colonization by OF is associated with reduced urinary oxalate excretion. Exposure to antibiotics may be an important factor contributing to variable rates of colonization. This is the first prospective study to evaluate the effect of antibiotics on OF colonization.

Design, setting, participants, & measurements: The effect of antibiotics on OF colonization was compared in 2 groups: a group receiving antibiotics for gastric infection with Helicobacter pylori (HP) and a group without HP that not receiving antibiotics. OF colonization in stool was detected by oxalate degradation at baseline and after 1 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* undergoing upper endoscopy
* H. pylori present or absent on gastric histology
* stool positive for Oxalobacter formigenes

Exclusion Criteria:

* unable to consent
* stool negative for Oxalobacter formigenes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing upper endoscopy for any indication and who would have determination of presence or absence of H. pylori. Stool samples then positive for colonization with Oxalobacter formigenes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2003-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Principal Investigator — New York Harbor VA Medical Center